CLINICAL TRIAL: NCT00854724
Title: Puerarin (NPI-031G) Effects on Alcohol Drinking - A Natural Settings Study
Brief Title: Puerarin Effects on Alcohol Drinking
Acronym: PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, David M. Penetar, Psychologist, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P-000726; R44AA152200 (Other Grant/Funding Number: NIAAA)
Record Dates: First submitted 2009-02-27; First posted 2009-03-03 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — puerarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Puerarin (Active Comparator)
  Interventions: Drug: Puerarin, Placebo
- Placebo (Placebo Comparator): Sugar beet filler in capsule
  Interventions: Drug: Puerarin, Placebo

INTERVENTIONS:
Drug: Puerarin, Placebo — 400 mg, three times a day for 7 days
  Other Names: Puerarin: NPI-031G; Placebo: Sugar beet extract

SUMMARY:
This research is designed to assess the impact of pretreatment with puerarin (NPI-031G), a major ingredient in the plant kudzu, on alcohol drinking. Hypothesis: Short-term treatment with this compound will reduce alcohol self-administration in a simulated natural settings laboratory.

DETAILED DESCRIPTION:
Participants will have an opportunity to drink up to 6 beers, plus water and juice, during a 90 minute afternoon drinking session in our simulated apartment room laboratory. Drinking sessions will be conducted in the afternoon after participants take puerarin or placebo for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* moderate to heavy alcohol drinkers (20+ drinks per week)

Exclusion Criteria:

* alcohol dependence or treatment-seeking drinkers
* other drug abuse or dependence
* psychiatric disorders

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M. Penetar, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Behavioral Psychopharmacology Research Laboratory, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Lukas SE, Penetar D, Berko J, Vicens L, Palmer C, Mallya G, Macklin EA, Lee DY. An extract of the Chinese herbal root kudzu reduces alcohol drinking by heavy drinkers in a naturalistic setting. Alcohol Clin Exp Res. 2005 May;29(5):756-62. doi: 10.1097/01.alc.0000163499.64347.92. PMID 15897719

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Placebo, Then Puerarin | Puerarin, Then Placebo
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout
Arm/Group | Placebo, Then Puerarin | Puerarin, Then Placebo
Started | 7 | 7
Completed | 6 | 6
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Period: Second Intervention
Arm/Group | Placebo, Then Puerarin | Puerarin, Then Placebo
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Puerarin | Puerarin, Then Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.3 (2.9) | 24.5 (3.7) | 24.4 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Amount of Alcohol Consumed
Time Frame: During a 90 minute drinking session
Measure: Mean (Standard Error); unit: Number of drinks consumed
Arm/Group | Placebo, Then Puerarin | Puerarin, Then Placebo
Number analyzed (Participants) | 8 | 8
Number of drinks consumed | 3.46 (0.55) | 2.36 (0.41)

ADVERSE EVENTS:
Arm/Group | Placebo, Then Puerarin | Puerarin, Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo, Then Puerarin (N=8) | Puerarin, Then Placebo (N=8)
headache (General disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Urinary Tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Cheek Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Elevated Liver Enzymes (Hepatobiliary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes